CLINICAL TRIAL: NCT05949697
Title: A Prospective Study of the Dry Eye Drink by Bruder Healthcare That Evaluates Hydration and Subject's Assessment on Eye Dryness
Brief Title: A Prospective Study of the Dry Eye Drink That Evaluates Hydration and Subject's Assessment on Eye Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruder Healthcare (Industry)
Collaborators: CBCC Global Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MW230012
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
Keywords: Eye Dryness; Dry Eye Drink
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dry Eye Drink (Other)
  Interventions: Dietary Supplement: Dry Eye Drink

INTERVENTIONS:
Dietary Supplement: Dry Eye Drink — Dry Eye Drink is a dietary supplement containing electrolytes, vitamins and natural anti-inflammatories.

SUMMARY:
A study to assess the effect of the Dry Eye Drink on eye dryness

DETAILED DESCRIPTION:
This is a prospective, non-randomized, comparative study of the Dry Eye Drink by Bruder Healthcare that evaluates hydration and subject's assessment on eye dryness. Subjects will administer the Dry Eye Drink by adding one sachet of the Dry Eye Drink powder in 12 Oz of water.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects aged between 18 and 65 years (both limits inclusive).
* Subjects with symptomatic Dry Eye Syndrome confirmed at baseline in at least any one or both the eyes.
* Subjects with ≥ 310 mOsmol/L tear osmolarity.
* Subjects with ≥ 6 SPEED score.
* Subject willing to provide written informed consent and able to comply with protocol requirements.

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period.
* Have undergone mechanical treatment for meibomian gland dysfunction using thermal pulsation/expression (e.g., LipiFlow) or intense pulsed light (e.g., OptiLight) therapy within 6 months prior to the Screening/Baseline Visit
* Have a known hypersensitivity to any of the study product components
* Have undergone ocular surgery (e.g., cataract, corneal or refractive surgical procedure) within 6 months prior to the Screening/Baseline Visit
* Have evidence of clinically significant ocular trauma
* Have active ocular Herpes simplex or Herpes Zoster infection
* Have ocular inflammation (uveitis, iritis, scleritis, episcleritis, conjunctivitis or keratitis, with the exception of keratoconjunctivitis sicca) at the discretion of the investigator
* Have ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids. including hordeolum)
* Have severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Have eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis)
* Have an ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity)
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Participation in any clinical study within 30 days before the first administration of study product.
* Subjects who are illiterate and cannot complete the subject diary independently.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change on the SPEED score | Day 0 and Day 30
  Change on the subjects' perception of eye dryness from Baseline to end of treatment as assessed by Standard Patient Evaluation of Eye Dryness (SPEED) score

SECONDARY OUTCOMES:
Change in Tear Osmolarity | Day 0 and Day 30
  Change in Tear Osmolarity from Baseline to end of treatment
Change in MMP-9 levels | Day 0 and Day 30
  Change in MMP-9 levels from Baseline to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CBCC Global Research Site:001, Bakersfield, California, United States